CLINICAL TRIAL: NCT07076680
Title: Safety and Effectiveness in Patients With HR+/HER2- Advanced Breast Cancer: a Prospective, Noninterventional Real-world Study
Brief Title: A Real-World Study in Patients With HR+/HER2- Advanced Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Due to a strategic decision by the company, the study will not proceed, and no subjects have been enrolled to date.
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: RWS
Record Dates: First submitted 2025-06-17; First posted 2025-07-22 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Metastatic; HR+/HER2- Advanced Breast Cancer
Keywords: HR+/HER2- advanced breast cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endocrine therapy

SUMMARY:
The goal of this observational study is to learn about the safety and effectiveness of people with advanced breast cancer that is hormone receptor-positive (HR+), HER2-negative (HER2-).

Participants will:

Allow researchers to collect medical data during routine care

Be followed for signs of treatment effectiveness and any medical problems that happen while taking the drug

ELIGIBILITY:
Inclusion Criteria:

* 1. must have a histologically or cytologically confirmed diagnosis of breast cancer and evidence of locally advanced or metastatic disease that is not amenable to surgical resection.

  2. Women or men ≥ 18 years of age. 3. must be confirmed as HR+ and HER2- by local laboratory tests. Confirmation of this status can be done by a first visit tissue sample or a post-treatment sample (recent biopsy sample preferred if available).

  4. Testing to confirm ESR1 mutation positivity should be performed on tumor DNA taken from tissue samples or circulating tumor DNA (ctDNA) obtained from plasma samples using a well-validated assay. Accept the results of the central laboratory or local laboratory tests, and in the event of inconsistency between the two test results, the investigator determines whether enrollment is possible.

  5. previous treatment with at least one endocrine therapy, either as monotherapy or in combination with another drug, at an advanced stage.

  6. have a life expectancy greater than 3 months and normal organ function (as assessed by the investigator).

Exclusion Criteria:

- 1. Pregnant or lactating females. 2. Known difficulty tolerating oral medications, or the presence of conditions that would interfere with the absorption of oral medications or allergies to medications and their excipients.

3. Other conditions that the investigator considers inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adults with advanced or metastatic breast cancer that is hormone receptor-positive (HR+), HER2-negative (HER2-), and has an ESR1 gene mutation. Participants will be receiving elacestrant as part of routine clinical care. They may be receiving treatment at cancer centers or hospitals across multiple regions in China. Both premenopausal and postmenopausal individuals may be eligible, based on local clinical practice.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From first dose until 30 days after last dose or end of follow-up (approximately 6 to 12 months)
  The number and percentage of participants who experience any adverse event (AE) during treatment, regardless of severity or causality. Events will be coded using standard terminology (e.g., MedDRA).

SECONDARY OUTCOMES:
Incidence of Serious Adverse Events (SAEs) | From first dose until 30 days after last dose or end of follow-up
  The number and percentage of participants who experience any serious adverse event (SAE), defined per ICH-GCP and local regulatory standards.
Rate of Dose Modifications Due to Adverse Events | From Day 1 (first dose) through the end of treatment (up to 24 months)
  The number and percentage of participants who require dose reductions or interruptions due to treatment-related adverse events.
Rate of Discontinuation Due to Adverse Events | From Day 1 (first dose) through the end of treatment (up to 24 months)
  The number and percentage of participants who permanently stop treatment due to treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jianli Zhao, Doctor, Principal Investigator — Sun Yat-sen Memorial Hospital, Sun Yat-sen University, China
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No